CLINICAL TRIAL: NCT00001632
Title: Myocardial Ultrasonic Tissue Characterization in Patients With a Genetic Predisposition for the Development of Hypertrophic Cardiomyopathy
Brief Title: Investigation Into the Use of Ultrasound Technique in the Evaluation of Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970188; 97-H-0188
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-08

CONDITIONS: Healthy; Hypertrophic Cardiomyopathy; Left Ventricular Hypertrophy
Keywords: Hypertrophy; Integrated; Backscatter; Cyclic; Echocardiography; Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy, Left Ventricular; Hypertrophy

SUMMARY:
The human heart is divided into four chambers. One of the four chambers, the left ventricle, is the chamber mainly responsible for pumping blood out of the heart into the circulation. Hypertrophic cardiomyopathy is a genetically inherited disease causing an abnormal thickening of heart muscle, especially the muscle making up the left ventricle. When the left ventricle becomes abnormally large, it is called left ventricular hypertrophy (LVH).

Patients with HCM can be born with an enlarged left ventricle or they may develop the condition in childhood or adolescence, usually during the time when the body is rapidly growing. However, not all patients with the abnormal genes linked to HCM have the characteristic LVH.

Currently, it is impossible to tell if a patient with the genes for HCM will develop LVH.

A recently developed ultrasound tool called an integrated backscatter analysis (IBS), may allow researchers to determine those children who may later develop HCM and LVH. In order to test this, researchers plan to use IBS to study normal children with relatives diagnosed with HCM.

This study will compare the results of IBS done on normal children with relatives diagnosed with HCM , normal children, and children with evidence enlarged heart muscle (HCM).

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is a genetically inherited disease that is characterized by unexplained left ventricular hypertrophy (LVH) often associated with diastolic dysfunction and myocardial ischemia. In patients with HCM, LVH may be present at birth or it may develop during childhood and adolescence, usually during periods of rapid body growth. Currently, it is not possible to identify, using clinical or laboratory methods, those children who will develop LVH from among those with a genetic predisposition for the disease. It would therefore be beneficial to find predictors of LVH development in normal children who have family history of HCM. Integrated backscatter analysis (IBS) is a recently developed ultrasound tool that has been studied in patients with various cardiac diseases. Integrated myocardial backscatter has been shown to vary throughout the cardiac cycle in normal subjects, both pediatric and adult, with peak values occurring during diastole and minimum values in end systole. Several studies in both children and adults with HCM have shown a blunting of this variation in backscatter analysis. We hypothesize that patients with a genetic predisposition for HCM, but no echocardiographic evidence of the disease, may have a greater prevalence of alterations in integrated myocardial backscatter when compared to children without a family history of HCM. We therefore propose to examine the cyclic variation of integrated myocardial backscatter in children with a normal echocardiogram and a first-degree relative with HCM, and compare it with the results obtained in a group of normal children, as well as in a group of children with unequivocal echocardiographic evidence of HCM.

ELIGIBILITY:
INCLUSION CRITERIA:

Three groups of subjects (aged 1-15 years) will be studied: normal children, children with HCM, and children that are family members of patients with HCM, but do not themselves have any evidence of LVH.

CONTROL GROUP (NORM GROUP):

Normal children under the age of 15 who have a normal two-dimensional echocardiogram will be included in the study.

HYPERTROPHIC CARDIOMYOPATHY GROUP (HCM GROUP):

Patients with HCM (unexplained LVH on two-dimensional echocardiogram) under the age of 15 will be included.

Family History of Hypertrophic Cardiomyopathy Group (FHCM GROUP:

Normal children under the age of 15 who have a first-degree relative with HCM and a normal two-dimensional echocardiogram will be included.

EXCLUSION CRITERIA - CONTROL GROUP:

Exclusion criteria will be any historical or echocardiographic evidence of congenital or valvular heart disease or any form of cardiomyopathy.

EXCLUSION CRITERIA - HCM GROUP:

Exclusion criteria will be any evidence of congenital or valvular heart disease that may explain the presence of LVH.

EXCLUSION CRITERIA - FHCM GROUP:

Exclusion criteria will be any historical or echocardiographic evidence of congenital or valvular heart disease or other form of cardiomyopathy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 195
Dates: Start 1997-09; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Panza JA, Maron BJ. Relation of electrocardiographic abnormalities to evolving left ventricular hypertrophy in hypertrophic cardiomyopathy during childhood. Am J Cardiol. 1989 May 15;63(17):1258-65. doi: 10.1016/0002-9149(89)90187-2. PMID 2523641
- [Background] Miller JG, Perez JE, Sobel BE. Ultrasonic characterization of myocardium. Prog Cardiovasc Dis. 1985 Sep-Oct;28(2):85-110. doi: 10.1016/0033-0620(85)90020-9. No abstract available. PMID 3898225
- [Background] Vitale DF, Bonow RO, Calabro R, De Cristofaro M, Pacileo G, Caso P, Gerundo G, Bordini C, Losi MA, Rengo C, Rengo F. Myocardial ultrasonic tissue characterization in pediatric and adult patients with hypertrophic cardiomyopathy. Circulation. 1996 Dec 1;94(11):2826-30. doi: 10.1161/01.cir.94.11.2826. PMID 8941108